CLINICAL TRIAL: NCT00954629
Title: A 26 Week Placebo-controlled, Randomised, Double-blind, Parallel Group Study of the Efficacy and Safety of 2PX (Topical Strontium Chloride Hexahydrate) in Patients With Pain Due to Osteoarthritis of the Knee
Brief Title: A Study of the Efficacy and Safety of 2PX in Patients With Pain Due to Osteoarthritis of the Knee
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Smerud Medical Research International AS (Other)
Collaborators: SantoSolve AS (Industry)
Responsible Party: Thorfinn Ege, SantoSolve AS
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2PX-OA-03
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2010-03

CONDITIONS: Pain; Osteoarthritis
Keywords: Osteoarthritis; Pain; Knee
MeSH Terms: conditions — Pain; Osteoarthritis | interventions — strontium chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2PX (Experimental): Pain medication
  Interventions: Drug: strontium chloride hexahydrate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: strontium chloride hexahydrate — Topical solution to be applied twice daily for 26 weeks. Dosage of up till 4 ml per application.
  Arms: 2PX
Drug: Placebo — Topical solution to be applied twice daily for 26 weeks. Dosage up till 4ml per application.
  Arms: Placebo

SUMMARY:
The purpose of the study is to demonstrate the superiority of topically administered 2PX versus placebo (vehicle) control in terms of reduction in pain intensity and physical function.

DETAILED DESCRIPTION:
Primary objective: To demonstrate the superiority of topically administered 2PX versus placebo (vehicle) control in terms of reduction in pain intensity and physical function.

Secondary objectives: To prospectively measure other efficacy variables of topically administered 2PX in pain associated with osteoarthritis of the knee. To evaluate the safety and tolerability of topically administered 2PX.

ELIGIBILITY:
Inclusion Criteria:

* Male and female out-patients, 40 years or older.
* Subjects with documented OA of either one or both knees, as defined by the American College of Rheumatology (ACR) criteria ([Altman R, Asch E, Bloch D, et al (1986)]); i.e.knee pain and at least 3 out of the following 6 criteria in the target joint:

  * age >50 years
  * stiffness < 30 minutes
  * crepitus
  * bony tenderness
  * bony enlargement
  * no palpable warmth
* Radiological evidence of joint space narrowing in the target joint within 8 weeks prior to randomisation.
* Subjects with chronic, moderate to severe OA pain of the target knee:

  * present for more than 3 months, and for ≥ 20 days per month.
  * not controlled by, or intolerant of, oral NSAIDs, paracetamol, COX-2 inhibitors or weak opioids.
  * intensity at least moderate (i.e., actual WOMAC (pain questions 1-5) ≥ 10) on WOMAC OA index LK 3.1 at Visit 1, in the target knee, as recalled over the last 24 hours.

Exclusion Criteria:

* Subjects with any moderate to severe pain of other origin (e.g., fibromyalgia) which could confound assessment or self-evaluation of pain due to OA in the target knee.
* Subjects with any prosthesis fitted to the target knee.
* Subjects requiring treatment with any of the following agents/therapies within the specified periods or at any time during the study are excluded from participation:
* Any potent/strong opioid in the 4 weeks prior to randomisation (i.e., an opioid assumed to cause withdrawal symptoms upon abrupt discontinuation).
* Any topical or subcutaneously applied analgesic agents (e.g., capsaicin, NSAIDs) applied to the target knee within 7 days prior to randomisation.
* Any treatment which could alter the degree or nature of baseline OA pain planned within the study period.
* Intra-articular injections of corticosteroids in the target knee within the 2 months prior to randomisation.
* Intra-articular injections of hyaluronan in the target knee within 6 months prior to randomisation.
* Avascular necrosis in the target knee within 6 months prior to randomisation.
* Arthrosynthesis of the target knee within 12 months prior to randomisation.
* Arthroscopy of the target knee within 6 months prior to randomisation.
* Major trauma to the target knee within 6 months prior to randomisation.
* Infection in the target knee within 6 months prior to randomisation.
* Subjects who have previously been treated with 2PX.
* Subjects who have received an investigational drug or used an investigational device within the 30 days prior to randomisation.
* Subjects with a significant psychiatric disorder, in the opinion of the investigator, or subjects receiving strong anti-psychotic medication.
* Subjects with documented or suspected alcohol or drug abuse.
* Any ongoing or past history of malignant disease within the 5 years immediately prior to randomisation (with the exception of basal cell carcinoma).
* Pregnancy or ongoing lactation
* Female subjects of childbearing potential unwilling to use adequate contraceptive measures throughout the duration of the study. For the purpose of this study, adequate contraception is defined as:

  * oral, injected or implanted hormonal methods of contraception; OR
  * placement of an intrauterine device (IUD) or intrauterine system (IUS); OR
  * barrier methods of contraception: Condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository Note: Male sterilisation or abstinence are not acceptable methods of birth control and would preclude enrolment in the study.

Note: For post-menopausal women: less than 12 months since the last spontaneous menstrual bleeding will exclude the patient unless they are willing to utilise acceptable methods of contraception for the duration of the study.

* Male subjects able to conceive, who are unwilling to use barrier methods of contraception throughout the duration of the study
* Subjects unable to comply with the study assessments.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
The difference between the active and placebo group in the change from Baseline to the assessment after 26 weeks of treatment in the actual WOMAC Osteoarthritis Index LK 3.1 subscale score for pain and physical function. | 26 weeks

SECONDARY OUTCOMES:
WOMAC Osteoarthritis Index LK 3.1; total and non-pain subscales: | At Screening, Baseline, Weeks 2, 4, 12, 26 and 27.
Pain intensity will be assessed by asking the question 'What is the level of pain in your target knee right now? | Daily
Patient Global Impression of Change (PGIC) | At weeks 12 and 26
Clinician Global Impression of Change (CGIC) | At weeks 12 and 26
Use of rescue medication: The number of paracetamol tablets used each day will be recorded. | Daily
Incidence of Disease Flares: The number and extent of flares in osteoarthritis pain of the target knee between active and placebo groups during the course of treatment. | At weeks 2, 4, 12, 26, and 27

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Ratcliffe, MD, Principal Investigator — MAC Neuroscience centre in Blackpool, United Kingdom
Locations (14):
- Finland (3):
  - Site in Helsinki, Helsinki
  - Site at Kuopio, Kuopio
  - Site in Turku, Turku
- Poland (3):
  - Site in Bialystok, Bialystok
  - Site in Kraków, Krakow
  - Site in Warszawa, Warsaw
- Site in St-Petersburg, Saint Petersburg, Russia
- United Kingdom (7):
  - Site in Blackpool, Blackpool
  - Site in Bolton, Bolton
  - Site in Bradford, Bradford
  - Site in Manchester, Manchester
  - Site at Cheadle Hulme, Stockport
  - Site at Heald Green, Stockport
  - Site at Heaton Moor, Stockport